CLINICAL TRIAL: NCT04385758
Title: Community Paramedicine Program to Improve Diabetes Care Quality, Equity, and Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rozalina G. McCoy, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-001011
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Diabetes; Diabetes Mellitus
Keywords: Community paramedicine; Diabetes mellitus; Diabetes distress
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes-REM Program (Experimental)
  Interventions: Other: Diabetes-REM Program

INTERVENTIONS:
Other: Diabetes-REM Program — A comprehensive community paramedicine management program designed to support adults with uncontrolled diabetes and a recent emergency department visit or hospitalization

SUMMARY:
The purpose of this study is evaluate the effectiveness of Diabetes-REM (Rescue, Engagement, and Management), a comprehensive community paramedic (CP) program to support adults in Southeast Minnesota (Mower, Freeborn, and Olmsted counties) and Northwest Wisconsin (Barron, Rusk, and Dunn) who have uncontrolled diabetes (HbA1c ≥ 9%) and have experienced an emergency department (ED) visit or hospitalization for any cause in the prior 6 months.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Most recent hemoglobin A1c ≥ 9% within the last 2 years.
* Age ≥ 18 years old.
* Type 1 or type 2 diabetes.
* Paneled to a Mayo Clinic or Mayo Clinic Health System practice.
* Able to provide informed consent.
* Proficient in English.
* Community-dwelling.
* Live in Southeast Minnesota (Mower, Freeborn, or Olmsted counties) or Northwest Wisconsin (Barron, Rusk, or Dunn counties).

Inclusion Criteria (Paramedics):

•Community Paramedics who delivered the Diabetes-REM intervention.

Exclusion Criteria:

* Cognitive impairment precluding informed consent.
* Lack of conversational English skills.
* Resident of a long-term care facility.
* Enrolled in hospice.
* Enrolled in a care coordination or disease management program.
* Advanced or terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Diabetes Distress (using DDS) | 1 month
  The level of diabetes-related distress that is expressed by patient participants using the Diabetes Distress Scale (the DDS contains 17 questions, with responses ranging from "Not a Problem" (1) to "A Very Serious Problem" (6). Total scores use the sum of all responses divided by 17, with a mean item score of 3 or higher (moderate distress) indicating distress worthy of clinical attention.)

SECONDARY OUTCOMES:
Diabetes Distress (using DDS) | 4 months
  The level of diabetes-related distress that is expressed by patient participants using the Diabetes Distress Scale (the DDS contains 17 questions, with responses ranging from "Not a Problem" (1) to "A Very Serious Problem" (6). Total scores use the sum of all responses divided by 17, with a mean item score of 3 or higher (moderate distress) indicating distress worthy of clinical attention.)
Confidence in Diabetes Self-Management (using DSMQ) | 1 and 4 months
  The level of confidence patient participants express in managing their diabetes using the Diabetes Self-Management Questionnaire (DSMQ)
Health-Related Quality of Life (using EQ-5D) | 1 and 4 months
  Patients participants' self-reported health-related quality of life using the EuroQol 5-D (also known as EQ-5D; an instrument for measuring quality of life)
Self-Reported Hypoglycemia and Hyperglycemia | 1 and 4 months
  Incidences of hypoglycemia (blood glucose <70 mg/dL and <54 mg/dL) and hyperglycemia (blood glucose ≥250 mg/dL) as reported by patient participants

CONTACTS AND LOCATIONS:
Overall Officials: Rozalina McCoy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juntunen MB, Liedl CP, Carlson PN, Myers LA, Stickler ZR, Ryan Schultz JA, Meilander AK, Behnken E, Lampman MA, Rogerson MC, Fischer KM, McCoy RG. Diabetes Rescue, Engagement and Management (D-REM): rationale and design of a pragmatic clinical trial of a community paramedicine programme to improve diabetes care. BMJ Open. 2022 Apr 21;12(4):e057224. doi: 10.1136/bmjopen-2021-057224. PMID 35450906
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials